CLINICAL TRIAL: NCT04905407
Title: Tamibarotene in Combination With Venetoclax and Azacitidine in Previously Untreated Adult Patients Selected for RARA-positive AML Who Are Ineligible for Standard Induction Therapy
Brief Title: Tamibarotene Plus Venetoclax/Azacitidine in Participants With Newly Diagnosed Acute Myeloid Leukemia (AML)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: As per sponsor decision, the study was terminated.
Sponsor: Syros Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SY-1425-202
Record Dates: First submitted 2021-05-24; First posted 2021-05-27 (Actual); Results first posted 2025-02-24 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2025-01

CONDITIONS: Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — tamibarotene; venetoclax; Azacitidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Part 1: Tamibarotene/Venetoclax/Azacitidine (Experimental): Participants will receive the tamibarotene/venetoclax/azacitidine triplet combination as follows: Azacitidine (intravenously or subcutaneously) at 75 milligrams (mg)/square meter (m^2) once daily, on Days 1 through 7 of each 28-day therapy cycle (per VIDAZA USPI). Alternative dosing of azacitidine (Days 1 through 5, 8, and 9) will be permitted throughout the study.
  Venetoclax (orally) daily on Days 1 through 28 per standard of care. Standard of care daily dosing is 100 mg on Day 1, 200 mg on Day 2, and 400 mg on Day 3 and beyond.
  Tamibarotene 6 mg twice daily (BID) orally, on Days 8 through 28 of each 28-day therapy cycle. Tamibarotene will only be administered to participants who have been confirmed as RARA-positive.
  Interventions: Drug: Tamibarotene; Drug: Venetoclax; Drug: Azacitidine
- Part 2: Tamibarotene/Venetoclax/Azacitidine (Experimental): Participants will receive the tamibarotene/venetoclax/azacitidine triplet combination at the dose and regimen selected in Part 1.
  Interventions: Drug: Tamibarotene; Drug: Venetoclax; Drug: Azacitidine
- Part 2: Venetoclax/Azacitidine (Active Comparator): Participants will receive the venetoclax/azacitidine combination at the dose and regimen selected in Part 1.
  Interventions: Drug: Venetoclax; Drug: Azacitidine
- Part 3: Tamibarotene/Venetoclax/Azacitidine (Experimental): Part 2 participants treated with venetoclax/azacitidine who experience progressive disease, relapse after initial CR or CRi response, or treatment failure may begin subsequent treatment in Part 3, where tamibarotene will be added to their regimen.
  Interventions: Drug: Tamibarotene; Drug: Venetoclax; Drug: Azacitidine

INTERVENTIONS:
Drug: Tamibarotene — Tamibarotene tablets will be administered per dose and schedule specified in the arm.
  Arms: Part 1: Tamibarotene/Venetoclax/Azacitidine; Part 2: Tamibarotene/Venetoclax/Azacitidine; Part 3: Tamibarotene/Venetoclax/Azacitidine
Drug: Venetoclax — Venetoclax tablets will be administered per dose and schedule specified in the arm.
  Other Names: Venclexta
Drug: Azacitidine — Azacitidine injection will be administered per dose and schedule specified in the arm.
  Other Names: Vidaza

SUMMARY:
Tamibarotene is being studied as a treatment for participants with a type of leukemia called acute myeloid leukemia, or AML for short. Tamibarotene is being studied as a treatment for participants with AML whose cancer has a specific genetic abnormality characterized by the overexpression of the retinoic acid receptor alpha (RARA) gene. This genetic profile is found in about 3 of every 10 people with AML.

During the trial, tamibarotene will be given with 2 other drugs that are already used together to treat people who have AML and who cannot start treatment with standard chemotherapy.

DETAILED DESCRIPTION:
This study consists of 3 parts. In Part 1, the safety, tolerability, and pharmacokinetic (PK) evaluation of tamibarotene/venetoclax/azacitidine combination will inform the appropriate tamibarotene dose to be combined with the standard of care (SOC) venetoclax/azacitidine in Part 2 and Part 3. In Part 2, participants will be randomized 1:1 to receive either tamibarotene/venetoclax/azacitidine or venetoclax/azacitidine to compare the clinical activity of the 2 combinations. In Part 3, tamibarotene will be added to the venetoclax/azacytidine regimen of a subset of Part 2 participants who experience progressive disease, relapse after initial complete remission (CR) or CR with incomplete blood count recovery (CRi) response, or treatment failure.

ELIGIBILITY:
Note: all inclusion/exclusion criteria should be met prior to the first dose of venetoclax/azacitidine on Cycle 1 Day 1 with the exception of the RARA-biomarker test result referenced in inclusion criterion 2, which should be positive by Cycle 1 Day 8 to continue treatment on study.

Inclusion Criteria:

* All participants must have obtained a blood sample for RARA biomarker investigational assay testing prior to starting treatment on Cycle 1 Day 1. The results of the investigational biomarker assay for all participants must be confirmed as RARA-positive by Cycle 1 Day 8 to enroll (Part 1) or to be randomized (Part 2) in the study.
* Participants must have newly diagnosed, previously untreated non-acute promyelocytic leukemia (APL) AML with a bone marrow or peripheral blood blast count ≥20% and must be unlikely to tolerate standard intensive chemotherapy at the time of Cycle 1 Day 1 Visit due to age, performance status, or comorbidities based on at least one of the following criteria:

  * age ≥75 years old, or
  * age <75 years old, with at least one of the following:

    * Eastern Cooperative Oncology Group (ECOG) performance status of 3
    * cardiac history of congestive heart failure (CHF) or documented ejection fraction (EF) ≤50%
    * pulmonary disease with diffusing capacity of the lungs for carbon monoxide (DLCO) ≤65% or forced expiratory volume in one second (FEV1) ≤65%
    * creatinine clearance ≥30 milliliters (mL)/minute (min) to <45 mL/min based on the Cockcroft-Gault glomerular filtration rate estimation
    * hepatic impairment with total bilirubin >1.5 to ≤3.0 * upper limit of normal (ULN)
    * any other comorbidity that the investigator judges to be incompatible with intensive chemotherapy, and reviewed and approved by the sponsor.

Exclusion Criteria:

* Participants have APL.
* Participants have known active central nervous system involvement with AML.
* Prior treatment (before Cycle 1 Day 1) for the diagnosis of AML, myelodysplastic syndromes (MDS), or antecedent hematologic malignancy with any hypomethylating agent, venetoclax, chemotherapy, or hematopoietic stem cell transplantation (HSCT), with the exception of prior treatment with hydroxyurea.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2021-08-26 (Actual); Primary Completion 2024-08-12 (Actual); Study Completion 2024-08-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Kelly Executive Medical Director, MD, Study Director — Syros Pharmaceuticals
Locations (28):
- United States (15):
  - City of Hope, Duarte, California
  - UCLA Medical Center Division of Hematology/Oncology, Los Angeles, California
  - University of Colorado, Denver, Colorado
  - Sarah Cannon Research Institute at Colorado Blood Cancer Institute, Denver, Colorado
  - Hartford HealthCare, Hartford, Connecticut
  - Northside, Atlanta, Georgia
  - University of Mississippi, Jackson, Mississippi
  - HCA Midwest Research Medical Center, Kansas City, Missouri
  - Atlantic Health, Morristown, New Jersey
  - Roswell Park Comprehensive Cancer Center, Buffalo, New York
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Novant Health, Charlotte, North Carolina
  - The Ohio State University James Cancer Hospital, Columbus, Ohio
  - Oregon Health & Science University, Portland, Oregon
- France (13):
  - CHU Lyon Sud, Pierre-Bénite, Pierre Benite
  - CHU Angers, Angers
  - CH de la Côte Basque, Bayonne
  - Hôpital Avicenne Hématologie Clinique, Bobigny
  - CHU de Caen Normandie, Caen
  - CHU Limoges, Limoges
  - CHU de Nantes - Hôtel Dieu, Nantes
  - Hôpital l'Archet- CHU de Nice, Nice
  - CHU de Bordeaux - Hôpital Haut-Lévèque, Pessac
  - CHU de Poitiers, Poitiers
  - Hôpital Saint-Louis, Vellefaux
  - Centre Hospitalier de Versailles, Versailles
  - Institut Gustave Roussy, Villejuif

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: As per sponsor decision, the study was terminated.
Groups:
- Part 1: Tamibarotene/Venetoclax/Azacitidine: Participants received tamibarotene/venetoclax/azacitidine triplet combination as follows: Azacitidine (intravenously or subcutaneously) at 75 milligrams (mg)/square meter (m^2) once daily, on Days 1 through 7 of each 28-day therapy cycle (per VIDAZA USPI). Alternative dosing of azacitidine (Days 1 through 5, 8, and 9) was permitted throughout the study.
  Venetoclax (orally) daily on Days 1 through 28 per standard of care. Standard of care daily dosing was 100 mg on Day 1, 200 mg on Day 2, and 400 mg on Day 3 and beyond.
  Tamibarotene 6 mg twice daily (BID) orally, on Days 8 through 28 of each 28-day therapy cycle. Tamibarotene was administered to participants who have been confirmed as retinoic acid receptor alpha (RARA)-positive.
- Part 2: Tamibarotene/Venetoclax/Azacitidine: Participants received tamibarotene/venetoclax/azacitidine triplet combination as follows: Azacitidine (intravenously or subcutaneously) at 75 mg/m^2 once daily, on Days 1 through 7 of each 28-day therapy cycle (per VIDAZA USPI). Alternative dosing of azacitidine (Days 1 through 5, 8, and 9) was permitted throughout the study.
  Venetoclax (orally) daily on Days 1 through 28 per standard of care. Standard of care daily dosing was 100 mg on Day 1, 200 mg on Day 2, and 400 mg on Day 3 and beyond.
  Tamibarotene 6 mg BID orally, on Days 8 through 28 of each 28-day therapy cycle.
- Part 2: Venetoclax/Azacitidine: Participants received venetoclax/azacitidine combination as follows: Azacitidine (intravenously or subcutaneously) at 75 mg/m^2 once daily, on Days 1 through 7 of each 28-day therapy cycle (per VIDAZA USPI). Alternative dosing of azacitidine (Days 1 through 5, 8, and 9) was permitted throughout the study.
  Venetoclax (orally) daily on Days 1 through 28 per standard of care. Standard of care daily dosing was 100 mg on Day 1, 200 mg on Day 2, and 400 mg on Day 3 and beyond.
- Part 3: Tamibarotene/Venetoclax/Azacitidine: Part 2 participants treated with venetoclax/azacitidine combination (Azacitidine (intravenously or subcutaneously) at 75 mg/m^2 once daily, on Days 1 through 7 of each 28-day therapy cycle (per VIDAZA USPI). Alternative dosing of azacitidine (Days 1 through 5, 8, and 9) was permitted throughout the study.
  Venetoclax (orally) daily on Days 1 through 28 per standard of care. Standard of care daily dosing was 100 mg on Day 1, 200 mg on Day 2, and 400 mg on Day 3 and beyond) who experienced progressive disease, relapse after initial Complete Remission (CR) or Complete Remission With Incomplete Hematologic Recovery (CRi) response, or treatment failure received subsequent treatment in Part 3, where tamibarotene (6 mg BID orally, on Days 8 through 28 of each 28-day therapy cycle) was added to their regimen.
Period: Part 1 and Part 2
Arm/Group | Part 1: Tamibarotene/Venetoclax/Azacitidine | Part 2: Tamibarotene/Venetoclax/Azacitidine | Part 2: Venetoclax/Azacitidine | Part 3: Tamibarotene/Venetoclax/Azacitidine
Started | 10 | 25 | 26 | 0
Received at Least 1 Dose of Study Drug | 10 | 25 | 26 | 0
Intent to Treat Analysis Set (Intent-to-Treat (ITT) Analysis Set included all participants who were randomized in Part 2. Treatment groups for this population were determined according to the treatment assignment at the time of randomization.) | 0 | 25 | 26 | 0
Safety Analysis Set (Safety Analysis Set included all randomized participants who had received any amount of study drug (tamibarotene, venetoclax, or azacitidine). Treatment groups for this population were determined according to the actual treatment the participants received. Participants who had only received venetoclax and/or azacitidine were assigned to the doublet treatment group (venetoclax/azacitidine combination).) | 10 | 24 | 27 | 0
Modified Intent-to-Treat (mITT) Analysis Set (Modified Intent-to-Treat (mITT) Analysis Set included all RARA-positive participants who were randomized in Part 2 and started dosing from Cycle 1 Day 1. Treatment groups for this population were determined according to the treatment assignment at the time of randomization.) | 0 | 25 | 26 | 0
Response Evaluable Population (Response evaluable set included all RARA-positive participants enrolled in Part 1 who had received any amount of study drug (tamibarotene, venetoclax, or azacitidine) and had either completed at least 1 response assessment or have discontinued treatment due to clinical progression/progressive disease prior to any response assessments.) | 9 | 0 | 0 | 0
Completed | 1 | 17 | 17 | 0
Not Completed | 9 | 8 | 9 | 0
Not completed — Withdrawal by Subject | 2 | 1 | 1 | 0
Not completed — Death | 7 | 7 | 7 | 0
Not completed — Other than specified | 0 | 0 | 1 | 0
Period: Part 3
Arm/Group | Part 1: Tamibarotene/Venetoclax/Azacitidine | Part 2: Tamibarotene/Venetoclax/Azacitidine | Part 2: Venetoclax/Azacitidine | Part 3: Tamibarotene/Venetoclax/Azacitidine
Started | 0 | 0 | 0 | 5
Received at Least 1 Dose of Study Drug | 0 | 0 | 0 | 5
Safety Analysis Set | 0 | 0 | 0 | 5
Completed | 0 | 0 | 0 | 3
Not Completed | 0 | 0 | 0 | 2
Not completed — Death | 0 | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Population: Part 1 and Part 3 safety population included all enrolled participants who had received any amount of study drug (tamibarotene, venetoclax, or azacitidine). Part 2 intent to treat (ITT) population included all participants who were randomized in Part 2. Treatment groups for this population were determined according to the treatment assignment at the time of randomization. Data of Part 3 participants is being reported separately.
Groups:
- Part 1: Tamibarotene/Venetoclax/Azacitidine: Participants received tamibarotene/venetoclax/azacitidine triplet combination as follows: Azacitidine (intravenously or subcutaneously) at 75 mg/m^2 once daily, on Days 1 through 7 of each 28-day therapy cycle (per VIDAZA USPI). Alternative dosing of azacitidine (Days 1 through 5, 8, and 9) was permitted throughout the study.
  Venetoclax (orally) daily on Days 1 through 28 per standard of care. Standard of care daily dosing was 100 mg on Day 1, 200 mg on Day 2, and 400 mg on Day 3 and beyond.
  Tamibarotene 6 mg BID orally, on Days 8 through 28 of each 28-day therapy cycle. Tamibarotene was administered to participants who have been confirmed as RARA-positive.
- Part 3: Tamibarotene/Venetoclax/Azacitidine: Part 2 participants treated with venetoclax/azacitidine combination (Azacitidine (intravenously or subcutaneously) at 75 mg/m^2 once daily, on Days 1 through 7 of each 28-day therapy cycle (per VIDAZA USPI). Alternative dosing of azacitidine (Days 1 through 5, 8, and 9) was permitted throughout the study.
  Venetoclax (orally) daily on Days 1 through 28 per standard of care. Standard of care daily dosing was 100 mg on Day 1, 200 mg on Day 2, and 400 mg on Day 3 and beyond) who experienced progressive disease, relapse after initial CR or CRi response, or treatment failure received subsequent treatment in Part 3, where tamibarotene (6 mg BID orally, on Days 8 through 28 of each 28-day therapy cycle) was added to their regimen.
- Total: Total of all reporting groups
Arm/Group | Part 1: Tamibarotene/Venetoclax/Azacitidine | Part 2: Tamibarotene/Venetoclax/Azacitidine | Part 2: Venetoclax/Azacitidine | Part 3: Tamibarotene/Venetoclax/Azacitidine | Total
Number analyzed (Participants) | 10 | 25 | 26 | 5 | 66
Age, Categorical [Count of Participants; unit: Participants] — Population: The baseline characteristics data of Part 3 participants are reported separately.
  Participants
    Part 1 and Part 2: number analyzed (Participants) | 10 | 25 | 26 | 0 | 61
    Part 1 and Part 2: <=18 years | 0 | 0 | 0 | 0 | 0
    Part 1 and Part 2: Between 18 and 65 years | 4 | 2 | 0 | 0 | 6
    Part 1 and Part 2: >=65 years | 6 | 23 | 26 | 0 | 55
    Part 3: number analyzed (Participants) | 0 | 0 | 0 | 5 | 5
    Part 3: <=18 years | 0 | 0 | 0 | 0 | 0
    Part 3: Between 18 and 65 years | 0 | 0 | 0 | 0 | 0
    Part 3: >=65 years | 0 | 0 | 0 | 5 | 5
Sex: Female, Male [Count of Participants; unit: Participants] — Population: The baseline characteristics data of Part 3 participants are reported separately.
  Participants
    Part 1 and Part 2: number analyzed (Participants) | 10 | 25 | 26 | 0 | 61
    Part 1 and Part 2: Female | 6 | 13 | 12 | 0 | 31
    Part 1 and Part 2: Male | 4 | 12 | 14 | 0 | 30
    Part 3: number analyzed (Participants) | 0 | 0 | 0 | 5 | 5
    Part 3: Female | 0 | 0 | 0 | 1 | 1
    Part 3: Male | 0 | 0 | 0 | 4 | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: The baseline characteristics data of Part 3 participants are reported separately.
  Participants
    Part 1 and Part 2: number analyzed (Participants) | 10 | 25 | 26 | 0 | 61
    Part 1 and Part 2: Hispanic or Latino | 0 | 0 | 0 | 0 | 0
    Part 1 and Part 2: Not Hispanic or Latino | 6 | 11 | 7 | 0 | 24
    Part 1 and Part 2: Unknown or Not Reported | 4 | 14 | 19 | 0 | 37
    Part 3: number analyzed (Participants) | 0 | 0 | 0 | 5 | 5
    Part 3: Hispanic or Latino | 0 | 0 | 0 | 0 | 0
    Part 3: Not Hispanic or Latino | 0 | 0 | 0 | 0 | 0
    Part 3: Unknown or Not Reported | 0 | 0 | 0 | 5 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: The baseline characteristics data of Part 3 participants are reported separately.
  Participants
    Part 1 and Part 2: number analyzed (Participants) | 10 | 25 | 26 | 0 | 61
    Part 1 and Part 2: American Indian or Alaska Native | 1 | 1 | 0 | 0 | 2
    Part 1 and Part 2: Asian | 0 | 0 | 0 | 0 | 0
    Part 1 and Part 2: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
    Part 1 and Part 2: Black or African American | 2 | 2 | 0 | 0 | 4
    Part 1 and Part 2: White | 4 | 8 | 7 | 0 | 19
    Part 1 and Part 2: More than one race | 0 | 0 | 0 | 0 | 0
    Part 1 and Part 2: Unknown or Not Reported | 3 | 14 | 19 | 0 | 36
    Part 3: number analyzed (Participants) | 0 | 0 | 0 | 5 | 5
    Part 3: American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
    Part 3: Asian | 0 | 0 | 0 | 0 | 0
    Part 3: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
    Part 3: Black or African American | 0 | 0 | 0 | 0 | 0
    Part 3: White | 0 | 0 | 0 | 0 | 0
    Part 3: More than one race | 0 | 0 | 0 | 0 | 0
    Part 3: Unknown or Not Reported | 0 | 0 | 0 | 5 | 5

OUTCOME MEASURES:

1. Primary Outcome: Part 1: Number of Participants With Treatment Emergent Adverse Events (TEAEs)
Description: An adverse event (AE) was defined as any untoward medical occurrence that developed or worsened in severity during the conduct of a clinical study and does not necessarily have a causal relationship to the study drug. A TEAE was any untoward medical occurrence associated with use of a study drug/study participation, whether or not considered related to study drug after first dose. TEAEs were defined as those adverse events AEs with onset after the first dose of study treatment or existing events that worsened after the first dose during the study up until the last dose of study treatment plus 30 days. A summary of serious and non-serious AEs regardless of causality is located in 'Reported Adverse Events module'.
Time Frame: Up to 3 years
Population: Part 1 Safety Analysis Set included all enrolled participants who received any amount of study treatment (tamibarotene, venetoclax, or azacitidine).
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Tamibarotene/Venetoclax/Azacitidine
Number analyzed (Participants) | 10
Participants | 10

2. Primary Outcome: Part 2: Complete Remission/Complete Remission With Incomplete Hematologic Recovery (CR/CRi) Rate
Description: CR/CRi rate was estimated by the percentage of participants who achieved complete Remission (CR) and/or CR with incomplete hematologic recovery (CRi),CR/CRi (as determined by the investigator). CR was defined as absolute neutrophil count ≥1,000/µL, platelets count ≥100,000/µL, bone marrow blasts <5% and absence of circulating blasts and blasts with auer rods; absence of extramedullary disease.CRi was defined as absolute neutrophil count <1,000/µL, platelets count <100,000/µL, bone marrow blasts <5% and all CR criteria met except either neutrophils or platelets not recovered.
Time Frame: Up to 3 years
Population: Part 2 mITT Analysis Set included all RARA-positive participants who were randomized in Part 2 and started dosing from Cycle 1 Day 1.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Part 2: Tamibarotene/Venetoclax/Azacitidine | Part 2: Venetoclax/Azacitidine
Number analyzed (Participants) | 25 | 26
Percentage of participants | 60.00 [38.7 to 78.9] | 69.23 [48.2 to 85.7]

3. Secondary Outcome: Part 1: Overall Response Rate (ORR)
Description: ORR: percentage of participants who achieved a overall response as comprised of CR(ANC ≥1,000/µL, platelets count (PC) ≥100,000/µL, bone marrow blasts <5% and absence of circulating blasts and blasts with auer rods;absence of extramedullary disease),CRi (ANC <1,000/µL, PC <100,000/µL, bone marrow blasts <5% and all CR criteria met except either neutrophils or platelets not recovered), CRh (ANC >500/µL, PC >500,000/µL, bone marrow blasts <5% and all CR criteria met except ANC and platelets with partial recovery of peripheral counts), morphologically leukemia-free state (bone marrow blasts <5%, absence of blasts with auer rods and <5% blasts in marrow sample with a count of at least 200 nucleated cells or cellularity ≥10%. Absence of EMD. No hematologic criteria required.), or PR was defined as ANC <1,000/µL, PC <100,000/µL, ≥50% decrease from baseline, with decrease to 5-25. ORR was calculated as ORR (%)=number of overall responders/number of participants in the Safety Population×100.
Time Frame: Up to 3 years
Population: Part 1 response evaluable population included all RARA-positive participants enrolled in Part 1 who had received any amount of study drug (tamibarotene, venetoclax, or azacitidine) and had either completed at least 1 response assessment or have discontinued treatment due to clinical progression/progressive disease prior to any response assessments.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Part 1: Tamibarotene/Venetoclax/Azacitidine
Number analyzed (Participants) | 9
Percentage of participants | 77.78 [40.0 to 97.2]

4. Secondary Outcome: Part 1: Plasma Concentration of Tamibarotene
Time Frame: Day 8 and 22 of Cycle 1, Day 15 of Cycles 2 and 3 (cycle length = 28 days)
Population: While blood samples were collected to derive data for the planned PK outcome measures, the study was terminated prior to that data being generated, analyzed, summarized, or made available by the study sponsor. Therefore, no PK data can be presented here.
Arm/Group | Part 1: Tamibarotene/Venetoclax/Azacitidine
Number analyzed (Participants) | 0

5. Secondary Outcome: Part 2: Number of Participants With Treatment Emergent Adverse Events
Description: An AE was defined as any untoward medical occurrence that developed or worsened in severity during the conduct of a clinical study and does not necessarily have a causal relationship to the study drug. A TEAE was any untoward medical occurrence associated with use of a study drug/study participation, whether or not considered related to study drug after first dose. TEAEs were defined as those adverse events AEs with onset after the first dose of study treatment or existing events that worsened after the first dose during the study up until the last dose of study treatment plus 30 days. A summary of serious and non-serious AEs regardless of causality is located in 'Reported Adverse Events module'.
Time Frame: Up to 3 years
Population: Part 2 safety population included all randomized participants who had received any amount of study drug (tamibarotene, venetoclax, or azacitidine).
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2: Tamibarotene/Venetoclax/Azacitidine | Part 2: Venetoclax/Azacitidine
Number analyzed (Participants) | 24 | 27
Participants | 24 | 24

6. Secondary Outcome: Part 2: Complete Remission (CR) Rate
Description: CR rate was estimated by the percentage of participants who achieved complete remission (as determined by the investigator). CR was defined as absolute neutrophil count ≥1,000/µL, platelets count ≥100,000/µL, bone marrow blasts <5% and absence of circulating blasts and blasts with auer rods; absence of extramedullary disease.
Time Frame: Up to 3 years
Population: Part 2 mITT population included all RARA-positive participants who were randomized in Part 2 and started dosing from Cycle 1 Day 1.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Part 2: Tamibarotene/Venetoclax/Azacitidine | Part 2: Venetoclax/Azacitidine
Number analyzed (Participants) | 25 | 26
Percentage of participants | 48.00 [27.8 to 68.7] | 57.69 [36.9 to 76.6]

7. Secondary Outcome: Part 2: Complete Remission/ Complete Remission With Partial Hematologic Recovery (CR/CRh) Rate
Description: CR/CRh rate was estimated by the percentage of participants who achieved complete Remission (CR) and/or CR with partial hematologic recovery (CRh),CR/CRh (as determined by the investigator). CR was defined as absolute neutrophil count ≥1,000/µL, platelets count ≥100,000/µL, bone marrow blasts <5% and absence of circulating blasts and blasts with auer rods; absence of extramedullary disease.CRh was defined as absolute neutrophil count >500/µL, platelets count >500,000/µL, bone marrow blasts <5% and all CR criteria met except ANC and platelets with partial recovery of peripheral counts.
Time Frame: Up to 3 years
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Part 2: Tamibarotene/Venetoclax/Azacitidine | Part 2: Venetoclax/Azacitidine
Number analyzed (Participants) | 25 | 26
Percentage of participants | 48.00 [32.2 to 75.6] | 57.69 [42.7 to 83.6]

8. Secondary Outcome: Part 2: Duration of Complete Remission
Description: Duration of CR was defined as duration from the date of first documented evidence of CR to the date of relapse of disease (as determined by the investigator), or death due to any cause, whichever occurred first. CR was defined as absolute neutrophil count ≥1,000/µL, platelets count ≥100,000/µL, bone marrow blasts <5% and absence of circulating blasts and blasts with auer rods; absence of extramedullary disease.
Time Frame: Up to 3 years
Population: Part 2 mITT population included all RARA-positive participants who were randomized in Part 2 and started dosing from Cycle 1 Day 1. Here, overall number of participants analyzed signifies those participants who were evaluable for this outcome measure.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Part 2: Tamibarotene/Venetoclax/Azacitidine | Part 2: Venetoclax/Azacitidine
Number analyzed (Participants) | 4 | 6
days | 293.0 [66.0 to NA] — The upper limit of 95% confidence interval (CI) could not be calculated due to smaller number of participants with an event. | 256.5 [56.0 to NA] — The upper limit of 95% CI could not be calculated due to smaller number of participants with an event.

9. Secondary Outcome: Part 2: Duration of CR/CRi
Description: Duration of CR/CRi was defined as duration from the date of first documented evidence of CR/CRi to the date of relapse of disease (as determined by the investigator), or death due to any cause, whichever occured first.CR was defined as absolute neutrophil count ≥1,000/µL, platelets count ≥100,000/µL, bone marrow blasts <5% and absence of circulating blasts and blasts with auer rods; absence of extramedullary disease.CRi was defined as absolute neutrophil count <1,000/µL, platelets count <100,000/µL, bone marrow blasts <5% and all CR criteria met except either neutrophils or platelets not recovered.
Time Frame: Up to 3 years
Population: as for outcome 8
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Part 2: Tamibarotene/Venetoclax/Azacitidine | Part 2: Venetoclax/Azacitidine
Number analyzed (Participants) | 5 | 8
days | 293.0 [66.0 to NA] — The upper limit of 95% CI could not be calculated due to smaller number of participants with an event. | 253.0 [56.0 to 263.0]

10. Secondary Outcome: Part 2: Duration of CR/CRh
Description: Duration of CR/CRh was defined as duration from the date of first documented evidence of CR/CRh to the date of relapse of disease (as determined by the investigator), or death due to any cause, whichever occured first. CR was defined as absolute neutrophil count ≥1,000/µL, platelets count ≥100,000/µL, bone marrow blasts <5% and absence of circulating blasts and blasts with auer rods; absence of extramedullary disease. CRh was defined as absolute neutrophil count >500/µL, platelets count >500,000/µL, bone marrow blasts <5% and all CR criteria met except ANC and platelets with partial recovery of peripheral counts.
Time Frame: Up to 3 years
Population: as for outcome 8
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Part 2: Tamibarotene/Venetoclax/Azacitidine | Part 2: Venetoclax/Azacitidine
Number analyzed (Participants) | 4 | 6
days | 293.0 [66.0 to NA] — The upper limit of 95% CI could not be calculated due to smaller number of participants with an event. | 256.5 [56.0 to NA] — The upper limit of 95% CI could not be calculated due to smaller number of participants with an event.

11. Secondary Outcome: Part 2: Time to Complete Response
Description: Time to CR was defined as the duration from the date of Cycle 1 Day 1 visit to the date of the first documented evidence of CR as determined by the investigator. CR was defined as absolute neutrophil count ≥1,000/µL, platelets count ≥100,000/µL, bone marrow blasts <5% and absence of circulating blasts and blasts with auer rods; absence of extramedullary disease.
Time Frame: Up to 3 years
Population: as for outcome 8
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Part 2: Tamibarotene/Venetoclax/Azacitidine | Part 2: Venetoclax/Azacitidine
Number analyzed (Participants) | 12 | 15
days | 21.0 [16.0 to 25.0] | 25.0 [19.0 to 43.0]

12. Secondary Outcome: Part 2: Time to CR/CRi
Description: Time to CR/CRi was defined as the duration from the date of Cycle 1 Day 1 Visit to the date of the first documented evidence of CR/CRi as determined by the investigator. CR was defined as absolute neutrophil count ≥1,000/µL, platelets count ≥100,000/µL, bone marrow blasts <5% and absence of circulating blasts and blasts with auer rods; absence of extramedullary disease.CRi was defined as absolute neutrophil count <1,000/µL, platelets count <100,000/µL, bone marrow blasts <5% and all CR criteria met except either neutrophils or platelets not recovered.
Time Frame: Up to 3 years
Population: as for outcome 8
Measure: Median (Inter-Quartile Range); unit: days
Groups:
- Part 2: Venetoclax/Azacitidine: Participants received tamibarotene/venetoclax/azacitidine triplet combination as follows: Azacitidine (intravenously or subcutaneously) at 75 mg/m^2 once daily, on Days 1 through 7 of each 28-day therapy cycle (per VIDAZA USPI). Alternative dosing of azacitidine (Days 1 through 5, 8, and 9) was permitted throughout the study.
  Venetoclax (orally) daily on Days 1 through 28 per standard of care. Standard of care daily dosing was 100 mg on Day 1, 200 mg on Day 2, and 400 mg on Day 3 and beyond.
  Tamibarotene 6 mg BID orally, on Days 8 through 28 of each 28-day therapy cycle.
Arm/Group | Part 2: Tamibarotene/Venetoclax/Azacitidine | Part 2: Venetoclax/Azacitidine
Number analyzed (Participants) | 15 | 18
days | 21.0 [16.0 to 28.0] | 24.5 [19.0 to 36.0]

13. Secondary Outcome: Part 2: Time to CR/CRh
Description: Time to CR/CRh was defined as the duration from the date of Cycle 1 Day 1 Visit to the date of the first documented evidence of CR/CRh as determined by the investigator. CR was defined as absolute neutrophil count ≥1,000/µL, platelets count ≥100,000/µL, bone marrow blasts <5% and absence of circulating blasts and blasts with auer rods; absence of extramedullary disease. CRh was defined as absolute neutrophil count >500/µL, platelets count >500,000/µL, bone marrow blasts <5% and all CR criteria met except ANC and platelets with partial recovery of peripheral counts.
Time Frame: Up to 3 years
Population: as for outcome 8
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Part 2: Tamibarotene/Venetoclax/Azacitidine | Part 2: Venetoclax/Azacitidine
Number analyzed (Participants) | 12 | 15
days | 21.0 [16.0 to 25.0] | 25.0 [19.0 to 43.0]

14. Secondary Outcome: Part 2: Overall Response Rate
Description: as for outcome 3
Time Frame: Up to 3 years
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Part 2: Tamibarotene/Venetoclax/Azacitidine | Part 2: Venetoclax/Azacitidine
Number analyzed (Participants) | 25 | 26
Percentage of participants | 80.00 [59.3 to 93.2] | 73.08 [52.2 to 88.4]

ADVERSE EVENTS:
Time Frame: Up to 3 years
Description: Part 1 and Part 3 safety population included all enrolled participants who had received any amount of study drug (tamibarotene, venetoclax, or azacitidine). Part 2 safety population included all randomized participants who had received any amount of study drug (tamibarotene, venetoclax, or azacitidine).
Arm/Group | Part 1: Tamibarotene/Venetoclax/Azacitidine | Part 2: Tamibarotene/Venetoclax/Azacitidine | Part 2: Venetoclax/Azacitidine | Part 3: Tamibarotene/Venetoclax/Azacitidine
All-Cause Mortality (participants affected / at risk) | 7/10 | 7/24 | 7/27 | 2/5
Serious Adverse Events (participants affected / at risk) | 10/10 | 15/24 | 13/27 | 4/5
Other Adverse Events (participants affected / at risk) | 10/10 | 24/24 | 24/27 | 5/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1: Tamibarotene/Venetoclax/Azacitidine (N=10) | Part 2: Tamibarotene/Venetoclax/Azacitidine (N=24) | Part 2: Venetoclax/Azacitidine (N=27) | Part 3: Tamibarotene/Venetoclax/Azacitidine (N=5)
Febrile bone marrow aplasia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 1
Febrile bone marrow aplasia (Blood and lymphatic system disorders) | 0 | 1 | 1 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 2 | 5 | 6 | 2
Leukopenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 3 | 0 | 1 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 1 | 2 | 0
Cardiac failure (Cardiac disorders) | 0 | 1 | 1 | 0
Myocardial infarction (Cardiac disorders) | 0 | 0 | 1 | 0
Anal incontinence (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Volvulus (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Asthenia (General disorders) | 0 | 2 | 0 | 0
Fatigue (General disorders) | 0 | 1 | 1 | 0
General physical health deterioration (General disorders) | 0 | 1 | 0 | 0
Malaise (General disorders) | 0 | 1 | 0 | 0
Oedema peripheral (General disorders) | 0 | 1 | 1 | 0
Pyrexia (General disorders) | 0 | 0 | 2 | 0
Non-cardiac chest pain (General disorders) | 1 | 0 | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 0 | 1 | 0
Bronchopulmonary aspergillosis (Infections and infestations) | 1 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 1 | 0
COVID-19 (Infections and infestations) | 1 | 0 | 0 | 0
Dermo-hypodermitis (Infections and infestations) | 0 | 0 | 1 | 0
Device related infection (Infections and infestations) | 0 | 0 | 1 | 0
Diverticulitis (Infections and infestations) | 0 | 0 | 1 | 0
Enterocolitis infectious (Infections and infestations) | 1 | 0 | 0 | 0
Escherichia sepsis (Infections and infestations) | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 2 | 1 | 0
Pyelonephritis (Infections and infestations) | 0 | 1 | 0 | 0
Sepsis (Infections and infestations) | 2 | 2 | 1 | 0
Septic shock (Infections and infestations) | 0 | 0 | 1 | 0
Staphylococcal sepsis (Infections and infestations) | 0 | 1 | 1 | 0
Streptococcal bacteraemia (Infections and infestations) | 0 | 1 | 0 | 0
Urinary tract infection pseudomonal (Infections and infestations) | 0 | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 2 | 0 | 0
Femur fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Neutrophil count decreased (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Failure to thrive (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 2 | 0 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 2 | 2 | 0
Ischaemic stroke (Nervous system disorders) | 0 | 1 | 0 | 0
Metabolic encephalopathy (Nervous system disorders) | 0 | 1 | 0 | 0
Presyncope (Nervous system disorders) | 0 | 1 | 0 | 0
Sciatica (Nervous system disorders) | 0 | 0 | 1 | 0
Encephalopathy (Nervous system disorders) | 1 | 0 | 0 | 0
Confusional state (Psychiatric disorders) | 0 | 1 | 0 | 0
Disorientation (Psychiatric disorders) | 0 | 0 | 1 | 0
Mental status changes (Psychiatric disorders) | 1 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 2 | 1 | 0
Renal failure (Renal and urinary disorders) | 0 | 1 | 0 | 0
Urinary incontinence (Renal and urinary disorders) | 0 | 0 | 1 | 0
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Pyoderma gangrenosum (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 0 | 1 | 0
Hypotension (Vascular disorders) | 0 | 1 | 0 | 0
Phlebitis (Vascular disorders) | 0 | 0 | 1 | 0
Atrioventricular block complete (Cardiac disorders) | 1 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 1 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1: Tamibarotene/Venetoclax/Azacitidine (N=10) | Part 2: Tamibarotene/Venetoclax/Azacitidine (N=24) | Part 2: Venetoclax/Azacitidine (N=27) | Part 3: Tamibarotene/Venetoclax/Azacitidine (N=5)
Acute kidney injury (Renal and urinary disorders) | 1 | 0 | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 1 | 5 | 5 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 4 | 0 | 1
Asthenia (General disorders) | 1 | 3 | 4 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 1 | 0 | 0
COVID-19 (Infections and infestations) | 0 | 2 | 0 | 1
Cardiac failure (Cardiac disorders) | 0 | 1 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 1 | 0 | 0
Confusional state (Psychiatric disorders) | 1 | 2 | 2 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 1 | 0 | 0
Dermo-hypodermitis (Infections and infestations) | 0 | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 9 | 5 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 4 | 6 | 0
Failure to thrive (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 2 | 1 | 0
Fatigue (General disorders) | 2 | 4 | 4 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 1 | 1 | 0
General physical health deterioration (General disorders) | 0 | 0 | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 2 | 4 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 1 | 1 | 0
Hypotension (Vascular disorders) | 1 | 0 | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 2 | 1 | 0 | 1
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 2 | 0
Nausea (Gastrointestinal disorders) | 3 | 7 | 9 | 0
Neutropenia (Blood and lymphatic system disorders) | 2 | 5 | 8 | 2
Neutrophil count decreased (Investigations) | 2 | 5 | 3 | 0
Oedema peripheral (General disorders) | 3 | 6 | 2 | 0
Phlebitis (Vascular disorders) | 0 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 2 | 1 | 0 | 0
Pyrexia (General disorders) | 1 | 1 | 4 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Sciatica (Nervous system disorders) | 0 | 1 | 0 | 0
Sepsis (Infections and infestations) | 0 | 2 | 1 | 0
Urinary incontinence (Renal and urinary disorders) | 0 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 2 | 4 | 0
Abdominal distension (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 2 | 1 | 3 | 0
Abdominal pain lower (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Activated partial thromboplastin time prolonged (Investigations) | 0 | 1 | 0 | 0
Agitation (Psychiatric disorders) | 1 | 0 | 1 | 0
Alanine aminotransferase increased (Investigations) | 0 | 2 | 2 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1
Animal bite (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Anosmia (Nervous system disorders) | 0 | 0 | 1 | 0
Anxiety (Psychiatric disorders) | 3 | 0 | 1 | 0
Aphasia (Nervous system disorders) | 0 | 1 | 0 | 0
Appendicitis (Infections and infestations) | 0 | 0 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 2 | 2 | 0
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 5 | 2 | 0
Bacteraemia (Infections and infestations) | 0 | 1 | 0 | 0
Bacterial infection (Infections and infestations) | 0 | 0 | 1 | 0
Bacterial pyelonephritis (Infections and infestations) | 0 | 0 | 1 | 0
Blood bilirubin increased (Investigations) | 0 | 1 | 2 | 0
Blood creatinine increased (Investigations) | 2 | 2 | 1 | 0
Blood lactate dehydrogenase increased (Investigations) | 1 | 1 | 0 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 1 | 0
Brain contusion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Brain fog (Nervous system disorders) | 0 | 0 | 1 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 1
Bronchostenosis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Bundle branch block (Cardiac disorders) | 0 | 0 | 1 | 0
Cachexia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Candida infection (Infections and infestations) | 0 | 1 | 0 | 0
Catheter site erythema (General disorders) | 0 | 1 | 0 | 0
Catheter site irritation (General disorders) | 0 | 1 | 1 | 0
Catheter site pain (General disorders) | 0 | 2 | 0 | 0
Chest pain (General disorders) | 0 | 0 | 0 | 1
Chills (General disorders) | 0 | 2 | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 1 | 0
Chondrocalcinosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Chronic kidney disease (Renal and urinary disorders) | 0 | 1 | 0 | 0
Clostridium difficile infection (Infections and infestations) | 0 | 1 | 1 | 0
Colitis ischaemic (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 5 | 10 | 5 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 5 | 5 | 0
Cryptosporidiosis infection (Infections and infestations) | 0 | 0 | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 5 | 5 | 7 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 2 | 0 | 0
Depression (Psychiatric disorders) | 0 | 0 | 1 | 0
Device malfunction (Product Issues) | 0 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 1 | 1 | 5 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 2 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Dysgeusia (Nervous system disorders) | 0 | 3 | 3 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 3 | 1 | 0
Dysuria (Renal and urinary disorders) | 0 | 1 | 1 | 0
Ear discomfort (Ear and labyrinth disorders) | 0 | 0 | 1 | 0
Ecchymosis (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0
Electrocardiogram T wave abnormal (Investigations) | 0 | 1 | 0 | 0
Enterococcal bacteraemia (Infections and infestations) | 0 | 1 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0
Epstein-Barr virus infection reactivation (Infections and infestations) | 0 | 1 | 0 | 0
Erysipelas (Infections and infestations) | 0 | 0 | 1 | 0
Eye disorders (Vascular disorders) | 0 | 2 | 0 | 0
Facial pain (General disorders) | 0 | 1 | 0 | 0
Facial paralysis (Nervous system disorders) | 0 | 0 | 1 | 0
Flat affect (Psychiatric disorders) | 0 | 0 | 1 | 0
Flatulence (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Gait disturbance (General disorders) | 0 | 1 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 3 | 0
Generalised oedema (General disorders) | 0 | 0 | 2 | 0
Gingival hypertrophy (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Gout (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0
HCoV-OC43 infection (Infections and infestations) | 0 | 1 | 0 | 0
Haematoma (Vascular disorders) | 0 | 0 | 1 | 0
Haemophagocytic lymphohistiocytosis (Immune system disorders) | 0 | 1 | 0 | 0
Haemorrhage intracranial (Nervous system disorders) | 0 | 1 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 2 | 0
Headache (Nervous system disorders) | 2 | 3 | 3 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 1 | 1 | 0
Hyperphosphataemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0
Hypertension (Vascular disorders) | 2 | 1 | 1 | 0
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1 | 1 | 1 | 1
Hypervolaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Hypoacusis (Ear and labyrinth disorders) | 0 | 0 | 1 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 2 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 1 | 3 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 2 | 2 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 2 | 5 | 0
Influenza (Infections and infestations) | 0 | 1 | 0 | 0
Influenza like illness (General disorders) | 0 | 2 | 1 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Ingrowing nail (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Injection site pain (General disorders) | 0 | 1 | 1 | 0
Injection site reaction (General disorders) | 0 | 0 | 1 | 0
Insomnia (Psychiatric disorders) | 1 | 4 | 2 | 0
International normalised ratio increased (Investigations) | 1 | 1 | 0 | 0
Joint effusion (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Left ventricular failure (Cardiac disorders) | 0 | 0 | 1 | 0
Lip oedema (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Lymphocyte count decreased (Investigations) | 0 | 2 | 3 | 0
Malnutrition (Metabolism and nutrition disorders) | 1 | 1 | 1 | 0
Mastoid disorder (Ear and labyrinth disorders) | 0 | 1 | 0 | 0
Melaena (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Memory impairment (Nervous system disorders) | 0 | 1 | 1 | 0
Mouth haemorrhage (Gastrointestinal disorders) | 0 | 2 | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 2 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 3 | 2 | 0 | 1
Myopericarditis (Cardiac disorders) | 0 | 0 | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 1 | 0
Ocular discomfort (Vascular disorders) | 0 | 1 | 0 | 0
Odynophagia (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Oesophageal candidiasis (Infections and infestations) | 0 | 1 | 0 | 0
Oral candidiasis (Infections and infestations) | 0 | 0 | 1 | 0
Oral fungal infection (Infections and infestations) | 0 | 1 | 0 | 0
Oral herpes (Infections and infestations) | 0 | 0 | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 1 | 0
Orthostatic hypotension (Vascular disorders) | 0 | 1 | 1 | 0
Oxygen saturation decreased (Investigations) | 0 | 0 | 1 | 0
Pain (General disorders) | 1 | 1 | 2 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 2 | 1 | 0
Pancreatic cyst (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Pancytopenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 1 | 1 | 0
Paranasal sinus discomfort (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Pericardial effusion (Cardiac disorders) | 0 | 3 | 0 | 0
Pericarditis (Cardiac disorders) | 0 | 0 | 1 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 1 | 0 | 0
Petechiae (Skin and subcutaneous tissue disorders) | 1 | 2 | 1 | 0
Physical deconditioning (General disorders) | 0 | 2 | 1 | 0
Platelet count decreased (Investigations) | 3 | 5 | 3 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 2 | 2 | 0
Postoperative wound complication (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Postural orthostatic tachycardia syndrome (Cardiac disorders) | 0 | 1 | 0 | 0
Proctalgia (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 7 | 0 | 0
Pseudomonas infection (Infections and infestations) | 0 | 0 | 1 | 0
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Rales (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 2 | 1 | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 1 | 2 | 0
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 2 | 1 | 0
Retching (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Rhinitis (Infections and infestations) | 1 | 1 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0
Rhinovirus infection (Infections and infestations) | 0 | 0 | 1 | 0
Rhonchi (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Right atrial enlargement (Cardiac disorders) | 0 | 1 | 0 | 0
Right ventricular enlargement (Cardiac disorders) | 0 | 1 | 0 | 0
SARS-CoV-2 test positive (Investigations) | 0 | 0 | 1 | 0
Sarcopenia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Sialoadenitis (Infections and infestations) | 0 | 1 | 0 | 0
Sinus headache (Nervous system disorders) | 0 | 0 | 1 | 0
Sinus tachycardia (Cardiac disorders) | 1 | 1 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 1 | 0 | 0
Skin infection (Infections and infestations) | 1 | 1 | 0 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 1 | 2 | 1 | 0
Skin mass (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 0
Speech disorder (Nervous system disorders) | 0 | 0 | 1 | 0
Stomal hernia (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 3 | 0 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Supraventricular tachycardia (Cardiac disorders) | 0 | 1 | 0 | 0
Syncope (Nervous system disorders) | 0 | 1 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 2 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 3 | 1 | 3
Thrombosis (Vascular disorders) | 0 | 1 | 0 | 0
Tooth infection (Infections and infestations) | 0 | 0 | 1 | 0
Tremor (Nervous system disorders) | 1 | 2 | 0 | 0
Troponin increased (Investigations) | 1 | 0 | 1 | 0
Tumour lysis syndrome (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Upper respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Urinary hesitation (Renal and urinary disorders) | 0 | 0 | 1 | 0
Urinary retention (Renal and urinary disorders) | 0 | 1 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 1 | 1 | 0
Urosepsis (Infections and infestations) | 0 | 0 | 1 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 1 | 0
Vulvovaginal mycotic infection (Infections and infestations) | 0 | 1 | 0 | 0
Walking disability (Social circumstances) | 0 | 0 | 1 | 0
Weight decreased (Investigations) | 0 | 6 | 3 | 0
Weight increased (Investigations) | 0 | 2 | 3 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
White blood cell count decreased (Investigations) | 4 | 5 | 5 | 0
Wound (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Wound complication (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Wound infection (Infections and infestations) | 0 | 0 | 1 | 0
Nodal rhythm (Cardiac disorders) | 1 | 0 | 0 | 0
Deafness bilateral (Ear and labyrinth disorders) | 1 | 0 | 0 | 0
Diplopia (Eye disorders) | 1 | 0 | 0 | 0
Vision blurred (Eye disorders) | 1 | 1 | 0 | 0
Ocular discomfort (Eye disorders) | 0 | 1 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Catheter site related reaction (General disorders) | 1 | 0 | 0 | 0
Chest discomfort (General disorders) | 1 | 0 | 0 | 0
Injection site erythema (General disorders) | 1 | 0 | 0 | 0
Malaise (General disorders) | 1 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 1 | 0 | 0 | 0
Swelling face (General disorders) | 1 | 0 | 0 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Abscess oral (Infections and infestations) | 1 | 0 | 0 | 0
Escherichia urinary tract infection (Infections and infestations) | 1 | 0 | 0 | 0
Oral infection (Infections and infestations) | 1 | 0 | 0 | 0
Vascular device infection (Infections and infestations) | 1 | 0 | 0 | 0
Foot fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Blood urea increased (Investigations) | 1 | 0 | 0 | 0
Blood alkaline phosphatase increased (Investigations) | 1 | 0 | 0 | 0
Brain natriuretic peptide increased (Investigations) | 1 | 0 | 0 | 0
Electrocardiogram QT prolonged (Investigations) | 1 | 0 | 0 | 0
Respiratory syncytial virus test positive (Investigations) | 1 | 0 | 0 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hypernatraemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Neuropathy peripheral (Nervous system disorders) | 1 | 0 | 0 | 0
Presyncope (Nervous system disorders) | 1 | 0 | 0 | 0
Taste disorder (Nervous system disorders) | 1 | 0 | 0 | 0
Disorientation (Psychiatric disorders) | 1 | 0 | 0 | 0
Bladder dilatation (Renal and urinary disorders) | 1 | 0 | 0 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Note that the agreements are between the clinical sites and the Sponsor (or its agents), which restrict the clinical trial sites' rights to discuss or publish trial results after the trial is completed.

DOCUMENTS (2):
  • Study Protocol (2024-06-04): https://cdn.clinicaltrials.gov/large-docs/07/NCT04905407/Prot_000.pdf
  • Statistical Analysis Plan (2024-03-18): https://cdn.clinicaltrials.gov/large-docs/07/NCT04905407/SAP_001.pdf